CLINICAL TRIAL: NCT00461422
Title: Early Follicular GnRH Antagonist Supplementation Improves Fertilization and Embryo Cleavage Rates in IVF-ET GnRH Antagonist Cycles
Brief Title: Early Follicular Supplementation of Ganirelix in IVF 2004
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Collaborators: Organon (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: soltsman2004.CTIL
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-06

CONDITIONS: Infertility; IVF Treatment
Keywords: IVF; GnRH antagonist
MeSH Terms: conditions — Infertility | interventions — ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Standard Flexible antagonist protocol Addition of Ganirelix at first 3 days of the cycle
  Interventions: Drug: Ganirelix
- 2 (No Intervention): Standard Flexible antagonist protocol

INTERVENTIONS:
Drug: Ganirelix — sc injection of Ganirelix 0.25 mg per day
  Arms: 1

SUMMARY:
Our goal was to investigate whether early follicular supplementation of the GnRH antagonist to the flexible GnRH antagonist protocol, has a potential to improve IVF-ET clinical results

DETAILED DESCRIPTION:
GnRH antagonist offers many advantages when used in IVF-ET treatment, however, it is suspected to yield lower pregnancy rate when compared with the long GnRH agonist protocol.

Our goal was to investigate whether early follicular supplementation of the GnRH antagonist to the flexible GnRH antagonist protocol, has a potential to improve IVF-ET clinical results.

Consecutive patients are prospectively enrolled and randomly assigned to the study and control groups. Patients with low ovarian reserve or with uterine distortion are excluded from the study. Both groups are treated with recombinant FSH and the flexible GnRH antagonist protocol. Women in the study group are also treated with additional GnRH antagonist 0.25 mg/day on day 1, 2 and 3 of the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* infertility
* IVF candidate
* failure of previous IVF attempt

Exclusion Criteria:

* low ovarian reserve
* untreated distortion of uterine cavity
* medical contraindication for IVF treatment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
pregnancy rates | one cycle

SECONDARY OUTCOMES:
differences in hormonal levels | one cycle
differences in the basic treatment doses | one cycle
oocyte counts | one cycle
fertilization rate | one cycle
cleavage rate | one cycle

CONTACTS AND LOCATIONS:
Overall Officials: Yohnny S Younis, MD, Principal Investigator — The Ministry of Health, Israel
Locations (1):
- The Baruch Padeh medical center, Poriya, Tiberias, Israel